CLINICAL TRIAL: NCT02765490
Title: A Phase 2b, Multicenter, Randomized, Open-label Study to Investigate the Efficacy, Safety and Pharmacokinetics of Different Treatment Regimens of AL-335, Odalasvir, and Simeprevir in Treatment-naive and Treatment-experienced Subjects With Chronic Hepatitis C Virus Genotype 1, 2, 4, 5, and 6 Infection Without Cirrhosis
Brief Title: Efficacy and Safety of Combinations of AL-335, Odalasvir (ODV) and Simeprevir (SMV) in the Treatment of Chronic Hepatitis C Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108070; 64294178HPC2001 (Other: Janssen Research & Development, LLC); 2015-004200-38 (EudraCT Number)
Record Dates: First submitted 2016-05-05; First posted 2016-05-06 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; AL-335; Odalasvir; Simeprevir; ODV; SMV; ACH-3102; ACH-0143102; TMC435
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — adafosbuvir; odalasvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): AL-335 (800 mg), odalasvir (25 mg) and simeprevir (75 mg) once daily during 6 weeks.
  Interventions: Drug: AL-335; Drug: Odalasvir; Drug: Simeprevir
- Group B (Experimental): AL-335 (800 mg), odalasvir (25 mg) and simeprevir (75 mg) once daily during 8 weeks.
  Interventions: Drug: AL-335; Drug: Odalasvir; Drug: Simeprevir

INTERVENTIONS:
Drug: AL-335 — AL-335 800 mg (2*400) tablet will be administered once daily.
Drug: Odalasvir — Odalasvir 25 mg tablet will be administered once daily.
Drug: Simeprevir — Simeprevir 75 mg capsule will be administered once daily.

SUMMARY:
The purpose of this study is to evaluate the efficacy (proportion of subjects with SVR12), safety, tolerability and pharmacokinetics of an 8- and 6-week treatment regimen of AL-335, odalasvir (ODV) and simeprevir (SMV) in chronic HCV genotype 1, 2, 4, 5 or 6 infected subjects without cirrhosis.

DETAILED DESCRIPTION:
This is a Phase 2b multicenter study. The study will include a screening period of maximum 6 weeks, a treatment period of 6 or 8 weeks and a 24-weeks post-treatment follow-up period. The total study duration for each subject will be 36 to 38 weeks. This study investigates a 3 direct-acting antiviral agent (DAA) combination of AL-335 (HCV NS5B inhibitor), odalasvir (ODV) (a second generation HCV NS5A inhibitor) and simeprevir (SMV) (HCV NS3A4 protease inhibitor). The results of this study will enable the selection of treatment and duration to be further developed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with chronic hepatitis C virus (HCV) genotype 1, 2, 4, 5 or 6 infection
* Documented as treatment naive or experienced with a prior regimen consisting of Interferon (IFN) +/-Ribavirin (RBV) regimen without achieving sustained viral response
* Absence of cirrhosis
* Screening laboratory values within defined thresholds
* Must use specific contraceptive methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Co-infection with human immunodeficiency virus (HIV) or hepatitis B virus (HBV)
* Prior exposure to an HCV direct-acting antiviral agent (DAA), either in combination with pegylated interferon (PegIFN) or IFN-free
* Current or prior history of clinical hepatic decompensation
* History of clinically significant illness or any other medical disorder including cardiovascular conditions that may interfere with individual's treatment, assessment or compliance with the protocol
* Pregnant or a nursing female

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (28):
- Belgium (6):
  - Antwerp
  - Brussels
  - Edegem
  - Ghent
  - Kortrijik
  - Leuven
- Canada (6):
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Toronto, Ontario
  - Vaughan, Ontario
  - Monteral, Quebec
  - Montreal, Quebec
- Germany (5):
  - Berlin
  - Essen
  - Frankfurt
  - Hamburg
  - Leipzig
- Poland (5):
  - Lodz
  - Lublin
  - Mysłowice
  - Warsaw
  - Wroclaw
- Singapore, Singapore
- Spain (5):
  - Barcelona
  - Madrid
  - Málaga
  - Seville
  - Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks: Participants received AL-335 800 milligram (mg) (2*400) tablets, Odalasvir (ODV) 25 mg tablet, and Simeprevir (SMV) 75 mg capsule once daily (qd) orally in the morning for 6 weeks.
- Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks: Participants received AL-335 800 milligram (mg) (2*400) tablets, Odalasvir (ODV) 25 mg tablet, and Simeprevir (SMV) 75 mg capsule once daily (qd) orally in the morning for 8 weeks.
Period: Overall Study
Arm/Group | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks
Started | 183 | 182
Completed | 182 | 179
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks | Total
Number analyzed (Participants) | 183 | 182 | 365
Age, Continuous [Median (Full Range); unit: years] | 48 [19 to 69] | 49 [18 to 70] | 49 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 94 | 182
  Male | 95 | 88 | 183
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 14 | 23
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 10 | 19
  White | 161 | 153 | 314
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 46 | 35 | 81
  Canada | 33 | 30 | 63
  Germany | 15 | 17 | 32
  Spain | 27 | 31 | 58
  Italy | 24 | 29 | 53
  Poland | 32 | 29 | 61
  Singapore | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After End of Treatment (EOT) (SVR12)
Description: The SVR 12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) less than (<) lower limit of quantification (LLOQ; 15 international unit per milliliter [IU/mL]) detectable or undetectable 12 weeks after actual EOT.
Time Frame: Week 12 (Follow-Up Phase)
Population: Intent-To-Treat (ITT) population included all randomized participants who took at least 1 dose of the study drug [that is AL-335, Odalasvir (ODV) or Simeprevir (SMV)].
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks
Number analyzed (Participants) | 183 | 182
Percentage of Participants | 98.9 [96.1 to 99.9] | 97.8 [94.5 to 99.4]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After End of Treatment (SVR24)
Description: The SVR24 was defined as HCV RNA <LLOQ (detectable or undetectable) 24 weeks after End of Treatment (EOT).
Time Frame: Week 24 (Follow-Up Phase)
Population: ITT population included all randomized participants who took at least 1 dose of the study drug (i.e., AL-335, ODV or SMV). Last Observation Carried Forward (LOCF) method was used to impute the missing values.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks
Number analyzed (Participants) | 183 | 182
Percentage of Participants | 98.9 [96.1 to 99.9] | 97.3 [93.7 to 99.1]

3. Secondary Outcome: Number of Participants With Viral Relapse
Description: Viral Relapse: Participants who did not achieve SVR12, with HCV RNA <LLOQ at the EOT and confirmed HCV RNA greater than or equal to (>=) LLOQ during follow-up.
Time Frame: End of Treatment up to Week 24 (Follow up phase)
Population: ITT population included all randomized participants who took at least 1 dose of the study drug (i.e, AL-335, ODV or SMV).
Measure: Number; unit: Participants
Arm/Group | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks
Number analyzed (Participants) | 183 | 182
Participants | 1 | 4

4. Secondary Outcome: Number of Participants With Late Viral Relapse
Description: Late Viral Relapse: Participants who achieved SVR12 but had confirmed HCV RNA>=LLOQ afterwards during follow-up.
Time Frame: Up to Week 24 (Follow-up Phase)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks
Number analyzed (Participants) | 183 | 182
Participants | 0 | 1

5. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: On-treatment failure: Participants who did not achieve SVR12 and with confirmed HCV RNA>=LLOQ at the End of Treatment (EOT).
Time Frame: EOT up to Week 12 (Follow up Phase)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks
Number analyzed (Participants) | 183 | 182
Percentage of Participants | 0 | 0

6. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After End of Treatment (EOT)
Description: The SVR 4 was defined as participants were considered to have reached SVR4, if 4 weeks after the actual EOT, HCV RNA was <LLOQ (detectable or undetectable).
Time Frame: Week 4 (Follow-Up Phase)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks
Number analyzed (Participants) | 183 | 182
Percentage of Participants | 99.5 [97.0 to 100.0] | 98.4 [95.3 to 99.7]

ADVERSE EVENTS:
Time Frame: Screening up to Follow-up (Week 24)
Arm/Group | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks
All-Cause Mortality (participants affected / at risk) | 0/183 | 1/182
Serious Adverse Events (participants affected / at risk) | 7/183 | 4/182
Other Adverse Events (participants affected / at risk) | 83/183 | 85/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks (N=183) | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks (N=182)
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal Strangulation (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Infective Keratitis (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ivth Nerve Paresis (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 6 Weeks (N=183) | Arm B: AL-335 800 mg+ODV 25 mg+SMV 75 mg qd for 8 Weeks (N=182)
Diarrhoea (Gastrointestinal disorders) | 7 | 10
Nausea (Gastrointestinal disorders) | 13 | 5
Asthenia (General disorders) | 11 | 8
Fatigue (General disorders) | 27 | 21
Viral Upper Respiratory Tract Infection (Infections and infestations) | 13 | 19
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 13
Headache (Nervous system disorders) | 40 | 40
Insomnia (Psychiatric disorders) | 15 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT02765490/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT02765490/SAP_001.pdf